CLINICAL TRIAL: NCT06611098
Title: A Randomized, Controlled, Prospective and Multicenter Clinical Investigation Evaluating the Safety and Performance of ABIO3419 in Treating Knee Osteoarthritis.
Brief Title: New Treatment of Knee Osteoarthritis
Acronym: PIVHAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Symatese (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIN2403
Record Dates: First submitted 2024-09-23; First posted 2024-09-24 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthristis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABIO3419 (Experimental): Patients will be enrolled and randomised to receive ABIO3419 by intra-articular injection.
  Interventions: Device: Viscosupplements
- Synvisc (Active Comparator): Patients will be enrolled and randomised to receive Synvisc(r) by intra-articular injection.
  Interventions: Device: Viscosupplements

INTERVENTIONS:
Device: Viscosupplements — intra-articular injection

SUMMARY:
Osteoarthritis (OA) is a chronic degenerative joint disease characterized macroscopically by progressive damage of articular cartilage, joint space narrowing, subchondral bone remodelling, joint marginal osteophyte formation and synovitis. It is also characterized by a decrease of the concentration and molecular weight of the hyaluronic acid in the synovial fluid which ultimately leads to poor viscoelastic properties of synovial fluid and induction of proinflammatory pathways.

The intra-articular injection of viscosupplementation gel (mainly exogenous hyaluronic acid) represents one of the most used therapeutic strategies to treat osteoarthritis symptoms.

Several studies on knee Osteoarthritis, have shown that one or more weekly injection of viscosupplementation gel significantly relieves articular pain and ameliorates mobility and joint function for at least 6 months and more. Repeated courses of intra-articular injections are an effective and safe treatment for knee osteoarthritis symptoms.

Based on studies conducted on intra-articular viscosupplementation gels, the most common side effects expected are local transient and short-lived adverse events such as pain, swelling and arthralgia in the site of administration, which are fully reversible in the days following the injection. Furthermore, such local effects may occur in a minority of cases and are usually treated conservatively with ice, non-steroidal anti-inflammatory drugs, and relative rest.

DETAILED DESCRIPTION:
Pivotal clinical investigation, interventional, prospective, comparative, single-blinded, controlled with two arms, randomized, multicentre clinical trial designed to assess the performance and safety of ABIO3419 for the treatment of osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily given informed consent to investigation participation in writing encompassing consent to data recording and verification procedures.
* 2. Male and female subjects, aged 35 to 85 years (inclusive).
* 3. Subjects affected by knee osteoarthritis, as defined by American College of Rheumatology (ACR) clinical and radiographic criteria for OA of the knee, and meeting the following conditions:

  1. Non-severe Grade 2 to 3 osteoarthritis of the knee according to the Kellgren-Lawrence (KL) classification, confirmed by an extension face X-rays shot, supported by flexion face X-rays shot (optional) obtained within 6 months from the screening visit.
  2. Subjects suffering from OA symptoms of the target knee for at least 6 months prior to the screening visit.
* 4. Pain during walking on flat ground in the target knee of at least 40 mm and maximum 80 mm on a 0-100 mm VAS at the baseline visit (Visit 2).
* 5. Subjects in treatment failure of first line treatment with oral NSAIDS
* 6. Women of childbearing potential must have a negative urine pregnancy test prior to each injection.
* 7. Subject who is able to comply with the study requirements, at the Investigator's appreciation.

Exclusion Criteria:

- 1. Pregnant and breastfeeding women

* 2. Subject with bilateral OA of the knees is excluded if one of the following points is present on the non-targeted knee has:
* a visual analog scale (VAS) score greater than 30mm (> 30mm),
* a KL score is greater than 2 (>2)
* a dedicated pain relief medicine consumption.
* 3. Subject suffering from a severe or progressive disease or any other pathology which, according to the investigator, may interfere with evaluation of the results of the study: diabetes, autoimmune pathology, cardiac pathologies, hepatic deficiency, epilepsy, porphyria, rheumatoid arthritis or other systemic inflammatory process.
* 4. Subject who has a known history of severe multiple allergies, angioedema or anaphylactic shock according to the investigator opinion.
* 5. Subject with a known allergy or hypersensitivity to Hyaluronic Acid or bovine collagen.
* 6. Subject with a past history of severe streptococcal disease or an active streptococcus infection according to the investigator opinion.

  7. Subject with an infections, inflammation or skin diseases in the area of the injection site.

  8. Subject with a disorder that may impact wound healing such as connective tissue or immunosuppressive disorder.

  9. Subject having received chemotherapy agents, immunosuppressive medications within the past 3 months.

  10. Subject with bleeding disorders or subject having received medication (anti-platelet agents and anticoagulant) that will likely increase the risk of bleeding within the past 24 hours before injections.

  11. Subjects having received:
  1. Intra-articular steroid injections within 60 days of the baseline visit or during study participation. Oral corticosteroids within four weeks of the screening visit or during study participation.
  2. Chondroitinsulphate, glucosamine sulphate, diacereine, bisphosphonates or matrix metalloproteinase (MMP) inhibitors within 30 days prior to the baseline visit.
  3. Viscosupplementation of the target knee within 6 months prior to the baseline visit.
  4. Any kind of pain relief medicine and NSAIDs in the 24 hours prior to the baseline visit (V2).

     12. Subjects with a KL grade 4 patellofemoral osteoarthritis or subjects with a patellofemoral osteoarthritis KL grade higher than the femora-tibial one.

     13. Subjects with coxarthrosis. 14. Subjects having had any previous surgery in the target knee within 6 months prior to the screening visit, or any planned surgery in the target knee throughout the duration of the investigation.

     15. Subjects who have had arthroplasty at the target knee at any time. 16. Subjects having had diagnostic or surgical knee arthroscopy, or knee lavage in the target knee in the 6 months prior to the screening visit.

     17. Subjects that are candidate for knee replacement within the study period. 18. Subjects with body mass index (BMI) > 35 kg/m2. 19. Subjects with large intra-articular effusion of the target knee, venous or lymphatic stasis, inflammatory flare-up with various symptoms, local inflammation.

     20. Subjects with history of septic OA of any joint 21. Subjects with significant pain outside the target knee, including significant hip or back pain and with fibromyalgia.

     22. Subjects with clinically significant valgus/varus deformities, ligamentous laxity, or meniscal instability as assessed by the Investigator.

     23. Subjects with other musculoskeletal condition affecting the target knee that would impair assessment of the effectiveness in the target knee (e.g. Paget's disease of bone).

     24. Subjects with a current malignancy or having treatment for a malignancy, except non-melanoma skin cancer.

     25. Subjects with drug or alcohol abuse 26. Subject who is deprived of their freedom by administrative or legal decision.

     27. Subject living in a social or sanitary establishment. 28. Subject being in an exclusion period for a previous study or with a current or recent (<3 months) participation in another investigational study involving a drug or combined device with drug.

     29. Other condition preventing the subject to participate the study in the Investigator's opinion: subject deemed unreliable or incapable of understanding and complying with the study assessment or unrealistic expectations of treatment results.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the performance of ABIO3419 treatment versus the comparator in subjects at 3 months (V7) by assessing knee pain while walking on flat ground. | Month 3 after the last injection
  Assessment by the subjects itself of the pain at 3-months (V7) compared to the baseline (V2 before initial injection) using a Visual Analogue Scale (VAS_0-100mm).
  The statistical objective is to demonstrate the non-inferiority of ABIO3419 compared to the comparator.

SECONDARY OUTCOMES:
Evaluate the pain of the treated knee when walking on a flat ground throughout the study. | Before intra-articular injections at 1 week, 2 week and then at 2 week, 1 month and 6 month after the last injection
  Assessment by the subject itself of the pain compared to baseline (V2 before initial injection) using a Visual Analogue Scale (VAS_0-100mm), at 1 week (V3) and 2 weeks (V4) after the first injection, and then at 2 weeks (V5), 1 month (V6) and 6 months (V8) after the last injection.
Evaluate the overall safety throughout the study. | immediately after first injection, before and immediately after the injections at 1 week and 2 weeks, and then at 2 weeks, 1 month, 3 months and 6 months.
  Assessment by the investigators of the occurrence and severity of adverse events (AE) at each time visits: immediately after first injection (V2), before and immediately after the injections at 1 week (V3) and 2 weeks (V4), and then at 2 weeks (V5), 1 month (V6), 3 months (V7) and 6 months (V8).
Evaluate the device related complications rates throughout the study | Immediately after first injection, before and immediately after the injections at 1 week and 2 weeks, then at 2 weeks, 1 month, 3 months and 6 months after the last injection
  Assessment of the proportion of patient with at least one adverse device effect related to ABIO3419 (ADE) at each time visits: immediately after first injection (V2), before and immediately after the injections at 1 week (V3) and 2 weeks (V4), and then at 2 weeks (V5), 1 month (V6), 3 months (V7) and 6 months (V8) after the last injection.
Evaluate the general health status of the treated knee | Baseline (before initial injection), 1 week and 2 weeks after the first injection (before 2nd and 3rd injections) then 2 weeks, 1 month, 3 months and 6 months after the last injection.
  Assessment by the patient itself of the target-knee functional status using the Knee injury and Osteoarthritis Outcome Score (KOOS).
  The KOOS holds 42 items in 5 separately scored subscales: Pain (nine items); Symptoms (seven items); Function in daily living (17 items); Sport and Recreation Function (five items); Quality of Life (four items).
  A 5-grade Likert scale is used for all items scored from 0 (No Problems) to 4 (Extreme Problems).
  Each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Evaluate concomitant analgesic consumption of subjects | 1 week before the first injection, 1 week and 2 weeks after the first injection then 2 weeks, 1 month, 3 months and 6 months after the last injection
  Assessment of the average weekly consumption (number and dosage) of paracetamol and pain killer drugs by patients using a daily diary.
Evaluate ABIO3419 implant card readability and subject's understanding | Day 0 (after first injection)
  Assessment by subjects of the reading and understanding of ABIO3419 implant card after the first injection (V2) of ABIO3419 through a dedicated questionnaire
Evaluate investigators' satisfaction | Month 6
  Investigator assessment of overall satisfaction using a 6-month satisfaction questionnaire with four response possibilities for each item: Very satisfied / Satisfied / Neutral / Not satisfied.
Evaluate patients' satisfaction | Month 6
  Assessment by the subject of the overall satisfaction with a satisfaction questionnaire at 6 months with four response possibilities for each item: Very satisfied / Satisfied / Neutral / Not satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Kristaps KNOHENFELDS, Principal Investigator — Veselibas Centrs ZIN; Kalvis KRASTINS, Principal Investigator — Kalvja Krastina private practice; Manaa Zodelava, Principal Investigator — JSC "Evex Hospitals" Caraps Medline; Nano Emukhvari, Principal Investigator — LLC Israel-Georgian Medical Research Clinic Healthycore; Luba Lagvilava, Principal Investigator — Consilium Medulla Multiprofile Clinic; Ketevan Tsintsadze, Principal Investigator — LTD HEALTH
Locations (2):
- IRIS CRO, Mtskheta, Georgia, Georgia
- IRIS CRO, Riga, Latvia, Latvia

IPD SHARING:
Plan to Share IPD: No